CLINICAL TRIAL: NCT06965140
Title: An Explorative Study Investigating Differences on the Peristomal Skin Condition by Optical Coherence Tomography (OCT)
Brief Title: CP376 OCT Exploratory Skin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP376
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OCT scan + skin measurements abdominal and peristomal skin (Other): OCT scan + skin measurements abdominal and peristomal skin
  Interventions: Device: flat 1-piece open ostomy device

INTERVENTIONS:
Device: flat 1-piece open ostomy device — OCT scan and skin measurements of peristomal and abdominal skin

SUMMARY:
An explorative study investigating differences on the peristomal skin and the abdominal skin by Optimal Coherence (OCT) 12 subjects with an ileostomy using a flat 1-piece open ostomy device will be enrolled.

The investigation consists of 2 visits, a screening visit (V0) and a Baseline/test visit (V1). V1 will also terminate the study period .The total study duration will be extended to a maximum of approximately 1 week, depending on the interval between V0 and V1.

DETAILED DESCRIPTION:
An explorative study investigating differences on the peristomal skin and the abdominal skin by Optimal Coherence (OCT)

12 subjects with an ileostomy using a flat 1-piece open ostomy device will be enrolled. Subjects will use their standard of care ostomy device as intended and remove the device at the test visit.

The investigation consists of 2 visits, a screening visit (V0) and a Baseline/test visit (V1). V1 will also terminate the study period when the OCT scan and other skin measurements has been completed. The total study duration will be extended to a maximum of approximately 1 week, depending on the interval between V0 and V1.

The OCT scans and other skin measurements (TEWL, Hydration and Erythema measurements) will be performed on the skin when the ostomy device has been removed.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent
2. Is at least 18 years old
3. Has full legal capacity
4. Has an ileostomy
5. Is using a flat 1-piece open ostomy device
6. Have had the ileostomy for a year

Exclusion Criteria:

1. Is currently receiving or have within the past two months received radio-and/or chemotherapy
2. Is currently receiving or have within the past month received steroid treatment in the skin area used in the investigation, e.g. lotion, spray, injection or tablet
3. Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Thickness of the epidermal layer (assessed by OCT) | immediately after the OCT scan
  Scan of the peristomal skin

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Department of dermatology and venerology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided